CLINICAL TRIAL: NCT04219553
Title: Moving Antimicrobial Stewardship Into Community Pharmacy: A Pre-post Study of Acute Otitis Media Management
Brief Title: Antimicrobial Stewardship in Community Pharmacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Katherine Koroluk, Principal Investigator, University of Toronto
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 34327
Record Dates: First submitted 2017-11-05; First posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Otitis Media
Keywords: antimicrobial stewardship; pharmacies; community pharmacy services; anti-infective agents; drug utilization
MeSH Terms: conditions — Otitis Media | interventions — Antimicrobial Stewardship

STUDY DESIGN:
Intervention Model Description: Pre-post intervention study model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrospective group (Other): Comparator group (pre-intervention)
  Interventions: Other: Comparator (no intervention)
- Prospective group (Experimental): Study group (post-intervention)
  Interventions: Behavioral: Antimicrobial stewardship

INTERVENTIONS:
Behavioral: Antimicrobial stewardship — The multifaceted AMS intervention includes pharmacist education, a clinical decision support tool, a parent/guardian questionnaire, and individualized monthly audit and feedback with each pharmacist.
  Arms: Prospective group
Other: Comparator (no intervention) — No active intervention
  Arms: Retrospective group

SUMMARY:
Acute otitis media (AOM) is the most common indication for antibiotics for Canadian paediatric patients. As the gatekeepers of safe and effective prescription pharmacotherapy, community pharmacists are well positioned to influence and optimize antibiotic use. The purpose of this project is to develop, implement, and evaluate an antimicrobial stewardship program in the community pharmacy setting that aims to optimize antibiotic use for AOM. This nonrandomized pre-post study includes children aged 6 months to 12 years presenting with an antibiotic prescription for AOM at two community pharmacies in Toronto, Ontario. Participants are excluded if they exhibit signs/symptoms of mastoiditis, have an additional indication for systemic antibiotics, or parents/guardians cannot consent in English. The multifaceted AMS intervention includes pharmacist education, a clinical decision support tool, a parent/guardian questionnaire, and individualized monthly audit and feedback with each pharmacist. Prescriptions are reviewed and adapted by the pharmacist to optimize congruence with 2016 Canadian Paediatric Society AOM guidelines. The primary outcome is the percentage change in guideline congruence attributable to pharmacist intervention. This study will provide insight into the opportunities and barriers of developing large-scale antimicrobial stewardship programs for community pharmacies.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed systemic oral antibiotic therapy
* Antibiotics are indicated for the treatment of acute otitis media (AOM) as reported verbally or in writing by parent/guardian or prescriber

Exclusion Criteria:

* signs/symptoms of mastoiditis
* a diagnosis in addition to AOM for which systemic antibiotics are indicated
* parents/guardians cannot consent to the study in English

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 188 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Change in guideline congruence | Pre-post study intervention (comparison of two 4-6 month periods)
  % change in guideline congruence for overall antibiotic prescriptions as attributable to pharmacist intervention before and after study intervention

SECONDARY OUTCOMES:
Choice of antibiotic | Pre-post study intervention (comparison of two 4-6 month periods)
  % change in guideline congruence for choice of antibiotic before and after study intervention
Antibiotic dosing | Pre-post study intervention (comparison of two 4-6 month periods)
  % change in guideline congruence for antibiotic dose before and after study intervention
Antibiotic duration | Pre-post study intervention (comparison of two 4-6 month periods)
  % change in guideline congruence for antibiotic duration before and after study intervention
Acceptance of pharmacist recommendations | Post-intervention study arm (6 month period after start of intervention)
  The percentage of pharmacist recommendations that were accepted by prescribers and parents/guardians (descriptive statistic)
Balancing measure: resolution of AOM | 7-14 days after antibiotics were dispensed
  The percent of cases with symptom resolution for AOM

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Shoppers Drug Mart #500, Toronto, Ontario
  - Shoppers Drug Mart #994, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided